CLINICAL TRIAL: NCT03403166
Title: Metabolomics of the Dietary Approaches to Stop Hypertension (DASH) Dietary Pattern: A Secondary Data Analysis of the DASH Trial
Brief Title: Metabolomics of the Dietary Approaches to Stop Hypertension (DASH) Dietary Pattern
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00007383-2; K01DK107782 (NIH)
Record Dates: First submitted 2017-12-21; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Dietary Modification; Blood Pressure
MeSH Terms: interventions — Dietary Approaches To Stop Hypertension; Fruit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DASH diet: The DASH diet consisted of a high intake of fruits, vegetables, and low-fat dairy products. It included a wide range of sources of protein, such as meat, fish, poultry, nuts, and beans. Sugar-sweetened beverages, desserts, and red meat were restricted. In terms of nutrients, the DASH diet had a high amount of fiber and protein; low amounts of saturated fat, total fat, and cholesterol; and intake of potassium, magnesium, and calcium at levels close to the 75th percentile of U.S. consumption.
  Interventions: Behavioral: DASH diet
- Fruits and vegetables diet: Potassium and magnesium intake was similar to the 75th percentile of U.S. consumption. Fiber intake was high. The fruits and vegetables diet consisted of more fruits and vegetables and fewer snacks and desserts than the control diet, but otherwise was similar to the control diet.
  Interventions: Behavioral: Fruits and vegetables diet
- Control diet: For the control diet, macronutrient intake was similar to average U.S. consumption and intake of potassium, magnesium, and calcium were similar to the 25th percentile of U.S. consumption. Sodium intake was approximately 3 g/day in each diet.
  Interventions: Behavioral: Control diet

INTERVENTIONS:
Behavioral: DASH diet — Diet intervention
  Groups: DASH diet
Behavioral: Fruits and vegetables diet — Diet intervention
  Groups: Fruits and vegetables diet
Behavioral: Control diet — Diet intervention
  Groups: Control diet

SUMMARY:
The present record represents a secondary data analysis of the Dietary Approaches to Stop Hypertension (DASH) trial. Study data and specimens were accessed through the National Heart, Lung, and Blood Institute (NHLBI) Biologic Specimen and Data Repository Coordinating Center (BioLINCC). A global, untargeted, metabolomic profile was used to investigate biomarkers of the DASH dietary pattern as well as blood pressure change.

DETAILED DESCRIPTION:
The present study was conducted in order to: 1) quantify the metabolomic expression of the DASH dietary pattern; and 2) examine the relationship between metabolites that reflect the DASH dietary pattern and blood pressure change. This secondary data analysis leverages the completed DASH trial, a randomized feeding trial (N=459).

ELIGIBILITY:
Inclusion Criteria:

* Men and women with systolic blood pressure <160 mmHg and diastolic blood pressure 80-95 mmHg

Exclusion Criteria:

* Taking anti-hypertensive medication
* Poorly controlled diabetes mellitus
* Hyperlipidemia
* Cardiovascular event within the past 6 months
* Chronic disease that may interfere with participation
* Pregnancy or lactation
* Body mass index > 35 kg/m2
* Unwilling to stop taking vitamin or mineral supplements or antacids
* Kidney disease
* Consumption of >14 alcoholic beverages per week
* Did not consent to the use of biological specimens
* Did not attend the 8 week follow-up visit
* No serum specimen or insufficient volume of serum specimens in repository

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of men and women (aged 22 years and older) with systolic blood pressure <160 mmHg and diastolic blood pressure 80-95 mmHg who were not taking antihypertensive medication. The mean age was 44 years, about half were women, and approximately 2/3 were black or another race/ethnicity minority. The mean body mass index was 28 kg/m2 and mean blood pressure was 132/82 mmHg.
Sampling Method: Non-Probability Sample
Enrollment: 459 (Actual)
Dates: Start 1993-08 (Actual); Primary Completion 1997-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Serum metabolites | 8 week follow-up visit
  Metabolites were measured using a global, untargeted, metabolomic platform in serum specimens collected at the end of the 8 week diet intervention in the DASH trial. Reverse phase, untargeted ultrahigh-performance liquid chromatography tandem mass spectrometry quantification was used to measure metabolites. Peaks were quantified by calculating the area under the curve. Data were normalized to account for day-to-day instrumental variation. Compounds were identified by comparison to a library of purified standards or recurrent unknown entities and matches were determined based on retention time, mass-to-charge ratio, and chromatographic data. A relative measure of each metabolite (not absolute) is determined. The Metabolon (Durham, NC) platform quantifies over 1,000 compounds representing a broad range of metabolic compounds, including amino acids, carbohydrates, cofactors and vitamins, energy, lipids, nucleotides, peptides, and xenobiotics (chemicals, drugs, and food components).

SECONDARY OUTCOMES:
Blood pressure | 8 week follow-up visit
  The change in blood pressure was defined as the blood pressure level at the end of the 8 week diet intervention minus the blood pressure level at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Casey M. Rebholz, PhD, MS, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Derived] Kim H, Lichtenstein AH, Coresh J, Appel LJ, Rebholz CM. Serum proteins associated with LDL-C and non-HDL-C reduction in response to dietary interventions in the DASH and DASH-Sodium trials. Food Funct. 2025 Nov 10;16(22):8764-8772. doi: 10.1039/d5fo02593a. PMID 41143495
- [Derived] Kim H, Lichtenstein AH, Coresh J, Appel LJ, Rebholz CM. Serum protein responses to Dietary Approaches to Stop Hypertension (DASH) and DASH-Sodium trials and associations with blood pressure changes. J Hypertens. 2024 Oct 1;42(10):1823-1830. doi: 10.1097/HJH.0000000000003828. Epub 2024 Aug 1. PMID 39196693
- [Derived] Kim H, Appel LJ, Lichtenstein AH, Wong KE, Chatterjee N, Rhee EP, Rebholz CM. Metabolomic Profiles Associated With Blood Pressure Reduction in Response to the DASH and DASH-Sodium Dietary Interventions. Hypertension. 2023 Jul;80(7):1494-1506. doi: 10.1161/HYPERTENSIONAHA.123.20901. Epub 2023 May 10. PMID 37161796
- [Derived] Kim H, Lichtenstein AH, Ganz P, Du S, Tang O, Yu B, Chatterjee N, Appel LJ, Coresh J, Rebholz CM. Identification of Protein Biomarkers of the Dietary Approaches to Stop Hypertension Diet in Randomized Feeding Studies and Validation in an Observational Study. J Am Heart Assoc. 2023 Apr 4;12(7):e028821. doi: 10.1161/JAHA.122.028821. Epub 2023 Mar 28. PMID 36974735
- [Derived] Rebholz CM, Lichtenstein AH, Zheng Z, Appel LJ, Coresh J. Serum untargeted metabolomic profile of the Dietary Approaches to Stop Hypertension (DASH) dietary pattern. Am J Clin Nutr. 2018 Aug 1;108(2):243-255. doi: 10.1093/ajcn/nqy099. PMID 29917038